CLINICAL TRIAL: NCT01729559
Title: Venous Thromboembolic Prophylaxis After Major Trauma: A Randomized Controlled Trial of Three Times a Day Unfractionated Heparin Versus Twice a Day Enoxaparin
Brief Title: Venous Thromboembolic Prophylaxis After Trauma: Three Times a Day Unfractionated Heparin Versus Twice a Day Enoxaparin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-12-5973
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Venous Thromboembolic Disease; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: venous thromboembolic disease; deep vein thrombosis; pulmonary embolism; trauma; antithrombotic prophylaxis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Wounds and Injuries | interventions — Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5000 Units unfractionated Heparin Q 8 hr (Experimental): Low Dose Unfractionated Heparin (5000 Units) given every eight hours until primary or secondary outcome measure reached, discharge, or >30 days on trauma service.
  Interventions: Drug: 5000 Units unfractionated Heparin Q 8 hr
- 30mg enoxaparin Q12 hr (Active Comparator): Randomly assigned trauma patients to receive Low Molecular Weight Heparin (30mg enoxaparin) given subcutaneously every twelve hours until primary or secondary outcome measure reached, discharge, or >30 days on trauma service.
  Interventions: Drug: 30mg enoxaparin Q12 hr

INTERVENTIONS:
Drug: 5000 Units unfractionated Heparin Q 8 hr — Venous thromboembolic prophylaxis medication
  Other Names: LDUH
  Arms: 5000 Units unfractionated Heparin Q 8 hr
Drug: 30mg enoxaparin Q12 hr — Venous thromboembolic prophylaxis
  Other Names: Lovenox, LMWH, enoxaparin
  Arms: 30mg enoxaparin Q12 hr

SUMMARY:
The rate of venous thromboembolic events in trauma patients at high risk for deep vein thrombosis and pulmonary embolism receiving low dose unfractionated heparin every 8 hours will be equivalent or less than a similar group of patients given a standard every 12 hour dose of low molecular weight heparin.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a common and potentially life threatening complication of major trauma. The risk of developing deep vein thrombosis (DVT) following major trauma exceeds 50% unless adequate chemoprophylaxis is used. Recent national quality improvement initiatives, such as the Surgical Care Improvement Project (SCIP), mandate the risk stratification of hospitalized patients and the use of VTE prophylaxis based on the risk assessment. Low Molecular Weight Heparin (LMWH, enoxaparin) and Low Dose Unfractionated Heparin (LDUH) are commonly used alternatives for VTE chemoprophylaxis following major trauma. LMWH became favored in most trauma centers following a prospective randomized controlled trial comparing the two agents that demonstrated superior efficacy and equivalent safety of LMWH over a twice per day dosing of LDUH. The results of this study were largely responsible for practice guideline recommendation changes favoring the use of LMWH in trauma patients by both the American College of Chest Physicians (ACCP) and the Eastern Association for the Surgery of Trauma (EAST). , This landmark paper did not, however, utilize a three times a day (every 8 hours) dosing of LDUH for prophylaxis, which is the dosing schedule recommended by earlier trials. LDUH administered every 8 hours was demonstrated to have similar efficacy to LMWH in trauma patients in a recent retrospective study. These results call into question the validity of the conclusions of the 1996 study. Because LDUH is less expensive ($0.50/dose) than LMWH (Enoxaparin, $28/dose), similar effectiveness would imply a significant reduction in the cost of prophylaxis and increased value to patients, providers and accountable care organizations and tax-payers.

To validate this hypothesis the investigators propose to achieve the following study objectives:

1. Assess the degree of risk for VTE in each patient admitted to the trauma service
2. Determine the rate of VTE events in high risk trauma patients receiving either:

   * LMWH (30mg enoxaparin) given every twelve hours
   * LDUH (5000 Units unfractionated Heparin) given every eight hours.
3. Identify and quantify any adverse events associated with either treatment arm.
4. Compare the value of LMWH versus LDUH in the prophylactic treatment of VTE disease in trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Scripps Mercy Trauma Service
* ≥18 Years old
* Stratified to either Significant or Highest risk of VTE by ACCP guidelines

Exclusion Criteria:

* Estimated Injury Severity Score (ISS) ≤9
* Likely to be discharged before hospital day 7
* Systemic coagulopathy defined with an International Normalized Ratio (INR) of ≥1.2
* Body Mass Index (BMI) >40
* Likely to Survive for <7 Days
* Pregnancy
* Evidence of renal insufficiency (Cr ≥1.3)
* Delayed transfer to this facility (>24 hrs)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Shackford, MD, Principal Investigator — Scripps Mercy Hospital, Department of Trauma Surgery
Locations (1):
- Scripps Mercy Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 15, 2012 through September 15, 2014, consecutively admitted adult trauma patients were evaluated for eligibility for the study. Patients aged 18 years and older and at risk for Venous thromboembolic event (VTE) based on the American College of Chest Physicians guidelines were included.
Pre-assignment Details: Those with an estimated Injury Severity Score (ISS) equal to or less than 9, those expected to have a hospital length of stay less than seven days by reason of discharge or death, and prisoners were excluded.
Groups:
- 5000 Units Unfractionated Heparin Q 8 Hours: Low Dose Unfractionated Heparin (5000 Units) given every eight hours until primary or secondary outcome measure reached, discharge, or >30 days on trauma service.
  5000 Units unfractionated Heparin Q 8 hours: Venous thromboembolic prophylaxis medication. Patients were randomly assigned.
- 30mg Enoxaparin Q12 Hours: Randomly assigned trauma patients to receive Low Molecular Weight Heparin (30mg enoxaparin) given subcutaneously every twelve hours until primary or secondary outcome measure reached, discharge, or >30 days on trauma service.
  30mg enoxaparin Q12 hours: Venous thromboembolic prophylaxis
Period: Overall Study
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours
Started | 251 | 244
Completed | 220 | 216
Not Completed | 31 | 28
Not completed — Protocol Violation | 31 | 28

BASELINE CHARACTERISTICS:
Population: Basic demographic and clinical characteristics of trauma patients who met all inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours | Total
Number analyzed (Participants) | 220 | 216 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (21.2) | 46.4 (20.8) | 46.4 (21.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 64 | 124
  Male | 160 | 152 | 312
Region of Enrollment [Number; unit: participants]
  United States | 220 | 216 | 436
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (4.5) | 26.9 (5.2) | 26.5 (4.9)
Injury Severity Score [Median (Full Range); unit: units on a scale] — The Injury Severity Score (ISS) is an anatomical scoring system that provides an overall score for patients with multiple injuries. Each injury is assigned an Abbreviated Injury Scale (AIS) score allocated to one of six body regions (Head, Face, Chest, Abdomen, Extremities, External). The highest AIS scores among the three most severely injured body regions are squared and added together to produce the total ISS score. The ISS score ranges from 0 to 75. Each AIS score ranges from 1 to 6 (6 denotes an unsurvivable injury).
  units on a scale | 10 [1 to 50] | 9 [1 to 38] | 9 [1 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Deep Vein Thrombosis
Description: Patients will have a bilateral lower extremity duplex ultrasound performed by a registered vascular technologist twice per week if the patient is in the ICU, or once per week if the patient is on the trauma ward. All of the deep veins from the external iliac to and including the calf veins will be interrogated. Diagnosis of deep vein thrombosis (DVT) will be defined as absence of complete vein compressibility, presence of an echogenic thrombus within the vein, absence of color flow characteristics including lack of spontaneity, phasicity, pulsatility and augmentability as noted in the clinical practice guidelines of the American Thoracic Society. The vascular technologist and physician reading the ultrasound study will be blinded to the patient's enrollment status and randomization arm/medication group.
Time Frame: Within 30 days of hospital admission
Measure: Number; unit: percentage of patients
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours
Number analyzed (Participants) | 105 | 103
percentage of patients | 4.8 | 2.9
Statistical Analysis 1: Comparison: 5000 Units Unfractionated Heparin Q 8 Hours vs 30mg Enoxaparin Q12 Hours; Analysis was performed in a subset of patients who received at least one follow-up venous duplex ultrasound of the lower extremities; Test type: Non-Inferiority or Equivalence — A 10% noninferiority margin was selected based on a previous trial showing a difference in the incidence of DVT of 13% with the use of 30 mg of enoxaparin every 12 hours compared to 5,000 U of unfractionated heparin (UFH) every 12 hr. To achieve 90% power using an a priori margin of 10% with a one-sided alpha of 0.025, a total of 182 patients (91 in each arm) was required; p = 0.025, Chi-squared, Corrected — One-tailed test of the cumulative VTE incidence between treatment groups; Risk Difference (RD) = 6.5, 95% CI 2-sided [-2.9 to 15.8] — Unadjusted cumulative incidence values between the two treatment groups were subtracted to calculate the risk difference for VTE between groups. This difference was compared to the a priori 10% margin of difference using the 95% confidence interval
Statistical Analysis 2: Comparison: 5000 Units Unfractionated Heparin Q 8 Hours vs 30mg Enoxaparin Q12 Hours; Analysis was performed in the total sample of eligible patients and who received their assigned treatment (referred to as the "randomized treated sample"); Test type: Non-Inferiority or Equivalence — A 10% noninferiority margin was selected based on these data showing a difference in the incidence of DVT of 13% with the use of 30 mg of enoxaparin every 12 hours compared to 5,000 U of UFH every 12 hours. To achieve 90% power using an a priori margin of 10% with a one-sided alpha of 0.025, a total of 182 patients (91 in each arm) was required. This analysis was performed in the entire sample; p = 0.025, Chi-squared, Corrected — One-tailed test of the cumulative VTE incidence between treatment groups; Risk Difference (RD) = 3.1, 95% CI 2-sided [-1.6 to 7.7] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Pulmonary Embolus
Description: Patients with any or all of the following signs and symptoms suggestive of pulmonary embolism will have a CT angiogram (CTA) performed for diagnosis: Sudden onset of dyspnea, deterioration of existing dyspnea, decreased oxygen saturation (<92%), onset of pleuritic chest pain without another apparent cause, onset of tachycardia (>100), evidence of hypoxemia, hypocapnia, or respiratory alkalosis on arterial blood gas, or electrocardiographic changes reflecting right ventricular strain.
Time Frame: Within 30 days from admission to hospital
Measure: Number; unit: participants
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours
Number analyzed (Participants) | 105 | 103
participants | 1 | 0

3. Secondary Outcome: Bleeding Event
Description: Bleeding events will be classified by the Graafsma et al. severity of bleeding criteria (Major, Minor or No Bleeding). A major bleeding event will be defined as any overt bleeding following initiation of chemoprophylaxis associated with one or more of the following; a decrease in hemoglobin of ≥2 g/dL, bleeding leading to a transfusion of ≥2 units of packed red blood cells, a new retroperitoneal or intracranial bleed, or bleeding that warranted cessation of chemoprophylaxis treatment. Minor bleeding is defined as clinically evident bleeding not meeting criteria for major bleeding.
Time Frame: Within 30 days of admission to hospital
Measure: Number; unit: participants
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours
Number analyzed (Participants) | 105 | 103
participants | 2 | 3

4. Secondary Outcome: Heparin Induced Thrombocytopenia
Description: The possible occurrence of heparin induced thrombocytopenia (HIT) was investigated when any patient (in either low molecular weight heparin [LMWH] or low dose unfractionated heparin [LDUH] study arm) had a platelet count drop of ≥50% (from a baseline value at the time of initiation of VTE prophylaxis) between day 5 and 14 following initiation of chemoprophylaxis per American College of Chest Physicians (ACCP) guidelines.
Time Frame: Within 30 of admission to hospital
Measure: Number; unit: participants
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours
Number analyzed (Participants) | 105 | 103
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 30 days after admission.
Arm/Group | 5000 Units Unfractionated Heparin Q 8 Hours | 30mg Enoxaparin Q12 Hours
Serious Adverse Events (participants affected / at risk) | 3/220 | 1/216
Other Adverse Events (participants affected / at risk) | 3/220 | 5/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5000 Units Unfractionated Heparin Q 8 Hours (N=220) | 30mg Enoxaparin Q12 Hours (N=216)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Same as one of the outcomes.
Trauma-related mortality (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — Trauma-related in-hospital mortality within 30 days of admission following administration of treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5000 Units Unfractionated Heparin Q 8 Hours (N=220) | 30mg Enoxaparin Q12 Hours (N=216)
Bleeding events (Blood and lymphatic system disorders) | 3 (3) | 5 (5) — Minor or Major bleeding events

LIMITATIONS AND CAVEATS:
The lack of long-term follow-up to identify VTE events among patients who were either transferred or readmitted to other facilities with VTE-related events was not performed. Published risk estimates were inaccurate for our sample size calculation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No